CLINICAL TRIAL: NCT06964308
Title: Thoracoscopic Pleural Biopsy, Sohag University Hospital
Brief Title: Thoracoscopic Pleural Biopsy in Sohag University Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Osama Yehia, Resident, Department of cardiothoracic Surgery, Faculty of Medicine, Sohag University, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med--25-2-03MS
Record Dates: First submitted 2025-03-16; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracoscopic pleural biopsy (Other): This arm aims to evaluate the diagnostic efficacy, safety, and clinical outcomes of thoracoscopic pleural biopsy in the management of pleural diseases.
  Interventions: Procedure: thoracoscopic pleural biopsy.

INTERVENTIONS:
Procedure: thoracoscopic pleural biopsy. — This intervention aims to evaluate the diagnostic efficacy, safety, and clinical outcomes of thoracoscopic pleural biopsy in the management of pleural diseases.

SUMMARY:
This study aims to evaluate the diagnostic efficacy, safety, and clinical outcomes of thoracoscopic pleural biopsy in the management of pleural diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected pleural disease who have been referred for thoracoscopic pleural biopsy
* Age: Adults aged 18 years and older
* Patients should have undergone necessary preoperative evaluations, including imaging studies (e.g., chest X-ray, CT scan) that indicate a need for biopsy.

Exclusion Criteria:

* Contraindications to Thoracoscopic Biopsy: Patients with contraindications to thoracoscopic biopsy
* Infeasibility of Procedure: Patients with anatomical or physiological factors that make thoracoscopic biopsy technically unfeasible or unsafe (e.g., severe pleural adhesions or distorted anatomy).
* Alternative Diagnoses: Patients who have been definitively diagnosed with a condition that does not require thoracoscopic biopsy for further evaluation.
* Pregnancy: Pregnant women may be excluded due to potential risks to the fetus and the need for specific procedural considerations.
* Inability to Provide Consent: Patients who are unable to provide informed consent due to cognitive impairment, language barriers, or other reasons.
* Participation in Concurrent Studies: Patients currently participating in other clinical studies that could interfere with the outcomes of this study or affect their eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
early postoperative follow up for thoracoscopic pleural biopsy in the management of pleural diseases. | 3 days after procedure
  return to daily activity

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Solari E, Marcozzi C, Ottaviani C, Negrini D, Moriondo A. Draining the Pleural Space: Lymphatic Vessels Facing the Most Challenging Task. Biology (Basel). 2022 Mar 10;11(3):419. doi: 10.3390/biology11030419. PMID 35336793
- [Background] Yao X, Abd Hamid M, Sundaralingam A, Evans A, Karthikappallil R, Dong T, Rahman NM, Kanellakis NI. Clinical perspective and practices on pleural effusions in chronic systemic inflammatory diseases. Breathe (Sheff). 2020 Dec;16(4):200203. doi: 10.1183/20734735.0203-2020. PMID 33447289
- [Background] Shaikh F, Lentz RJ, Feller-Kopman D, Maldonado F. Medical thoracoscopy in the diagnosis of pleural disease: a guide for the clinician. Expert Rev Respir Med. 2020 Oct;14(10):987-1000. doi: 10.1080/17476348.2020.1788940. Epub 2020 Jul 12. PMID 32588676